CLINICAL TRIAL: NCT00715858
Title: A Pilot Study Comparing Inflammatory Biomarkers in Blood and CSF in Patients With Alzheimer's Disease and Age-Matched Controls
Brief Title: A Pilot Study of Inflammatory Markers in Alzheimer's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: William Molloy, McMaster University
Allocation: Non-Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: R07-63
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; dementia; inflammation; cytokine; biomarker; cerebrospinal fluid; serum; doxycycline; rifampin
MeSH Terms: conditions — Alzheimer Disease; Dementia; Inflammation | interventions — Doxycycline; Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 AD doxycycline + rifampin (Active Comparator): Participants with AD allocated to doxycycline 100 mg bid od and rifampin 300 mg od for 12 months
  Interventions: Drug: doxycycline; Drug: rifampin
- 2 AD doxycycline (Active Comparator)
  Interventions: Drug: doxycycline; Drug: placebo
- 3 AD rifampin (Active Comparator): Participants with AD allocated to rifampin 300 mg od od and placebo matched to doxycycline bid for 12 months
  Interventions: Drug: rifampin; Drug: placebo
- 4 AD placebo (Placebo Comparator): Participants with AD allocated to placebo matched to doxycycline and placebo matched to rifampin for 12 months
  Interventions: Drug: placebo
- 5 Control (No Intervention): Age-matched cognitively healthy participants (untreated)

INTERVENTIONS:
Drug: doxycycline — capsule, 100 mg, b.i.d., 12 months
  Other Names: Apo-doxy
  Arms: 1 AD doxycycline + rifampin; 2 AD doxycycline
Drug: rifampin — capsule, 300 mg, od, 12 months
  Other Names: rifampicin; Rofact; Rifadin
  Arms: 1 AD doxycycline + rifampin; 3 AD rifampin
Drug: placebo — placebo matched to rifampin; placebo matched to doxycycline
  Arms: 2 AD doxycycline; 3 AD rifampin; 4 AD placebo

SUMMARY:
The purpose of this study is to examine the cerebrospinal fluid (CSF) of patients with Alzheimer's disease for biomarkers of inflammation and their response to the antibiotics doxycycline and rifampin. The results of this preliminary analysis will be used in defining the direction of further research.

DETAILED DESCRIPTION:
Doxycycline and rifampicin are two antibiotics which may be useful in the treatment of Alzheimer's disease (AD). Besides their antimicrobial effects they may also decrease specific contributors to AD pathology including: 1. amyloid beta, 2. inflammatory mediators, 3. proteolytic enzymes, and 4. metal ions. Evidence indicates an inflammatory response in AD. This includes complement activation, elevated C-reactive protein (CRP), elevated pro-inflammatory cytokines (including IL-1-beta, IL-6, TNF-α, TGF-β, S100-β), chemokine alterations (IL-8, MIP-1-alpha, MIP-1-beta, MCP-1), and microglial activation. In our previous study of AD patients treated with combined doxycycline and rifampicin versus placebo, we demonstrated that antibiotic treatment significantly delayed progression of clinical impairment. Treatment also reduced blood CRP levels suggesting an anti-inflammatory role of these antibiotics. In this study we suggest analysis of biomarkers including both pro and anti-inflammatory cytokines TNF-alpha, IL-1beta, IL-4, IL-10,the chemokine MCP-1 and other inflammatory markers in both the cerebrospinal fluid (CSF) and blood from AD patients and age-matched controls.

AD patients are participants in a 12 month randomized clinical trial of doxycyline and rifampin or placebo (DARAD) for treatment of AD. Each patient is asked if they wish to contribute a sample of CSF and blood at baseline and at 12 months when treatment is completed. About half the patients are consenting to this. Since consent is given to the lumbar puncture before the double-blinded DARAD treatment is initiated, we expect the distribution of samples collected to be random among the four treatment groups. We will compare CSF biomarker levels among the four treatment groups. Ten age-matched healthy controls are also being asked to contribute CSF and blood samples for comparison. The controls are not participants in the DARAD trial.

We feel that this is an important pilot study to determine whether there are any differences in blood or CSF concentrations of commonly studied cytokines between AD patients and normal controls. As such, this study could contribute to the search for a diagnostic biomarker. Also, it could provide a solid foundation for future studies aimed at elucidating the effects of antibiotics on various biomarkers in the blood and CSF of AD patients. From this, we may be able to correlate previous findings that antibiotics delay progression of clinical outcome in AD with changes in blood or CSF biomarker levels.

ELIGIBILITY:
Inclusion Criteria:

* Giving informed consent to lumbar puncture
* Participation in the DARAD clinical trial which requires the following:
* diagnosis of probable Alzheimer's disease
* SMMSE 14-26 inclusive
* community-dwelling
* age 50 or greater
* caregiver to monitor study medication and report on ADLs, behaviour, etc.
* adequate English literacy to complete neuropsychological testing
* generally stable level of health

Exclusion Criteria:

* Contraindication to lumbar puncture
* DARAD exclusion criteria as follows:
* dementia due to other neurodegenerative diseases
* cognitive impairment due to head trauma, etc.
* stroke or significant cerebrovascular disease
* clinically significant cardiac disease such as recent MI, uncontrolled hypertension
* taking other anti-dementia treatments or investigational drugs
* allergy to doxycycline or rifampin
* significant psychiatric conditions like depression
* cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-08 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
IL-1beta | baseline and 12 months
TNF-alpha | baseline and 12 months
MCP-1 | baseline and 12 months
IL-4 | baseline and 12 month
IL-10 | baseline and 12 months

SECONDARY OUTCOMES:
Other inflammatory markers. | Baseline and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: D.William Molloy, MB, MRCPI, FRCPC, Study Chair — McMaster University; Brandon M Kucher, PhD, MD, Principal Investigator — McMaster University; Shucui Jiang, MD,PhD, Study Director — McMaster University; Michel P Rathbone, MB, PhD, Study Director — McMaster University
Locations (1):
- St.Peter's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Loeb MB, Molloy DW, Smieja M, Standish T, Goldsmith CH, Mahony J, Smith S, Borrie M, Decoteau E, Davidson W, McDougall A, Gnarpe J, O'DONNell M, Chernesky M. A randomized, controlled trial of doxycycline and rifampin for patients with Alzheimer's disease. J Am Geriatr Soc. 2004 Mar;52(3):381-7. doi: 10.1111/j.1532-5415.2004.52109.x. PMID 14962152
- See also: DARAD Study clinical trial registration on ISRCTN15039674. Details provided. — http://www.controlled-trials.com/